CLINICAL TRIAL: NCT04813978
Title: The Effect of Music Therapy on Preoperative Anxiety in Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, SURAJ NAMLEWAR, Principal investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SNAMLEWAR
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Anxiety; Music; Preoperative
Keywords: anxiety; music; preoperative
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Researcher provides music to one group and other group will not receive music. medical officer will assess anxiety by using Beck's Anxiety Inventory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (control) (No Intervention): Head phone will be placed and music will not be played, will get normal nursing care
- Group A (music intervention) (Experimental): For the interventional group, in addition to normal nursing care, patients will listen to instrumental relaxing music genre consist of pitch, rhythm and tone color for 30 minutes pre-operatively, using mp3 player and over-ear headphones to reduce outside interference, at a volume of the patient's preference.
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — For the interventional group, in addition to normal nursing care, patients will listen to instrumental relaxing music genre consist of pitch, rhythm and tone color for 30 minutes pre-operatively, using mp3 player and over-ear headphones to reduce outside interference, at a volume of the patient's preference.
  Arms: Group A (music intervention)

SUMMARY:
Anxiety is a common phenomenon among patients who are undergoing surgery. It is a condition characterized by stress, nervousness, fear, unpleasant feeling, and higher activity of Autonomic Nervous System. The current studies demonstrated that listening to music, reduces anxiety levels.

DETAILED DESCRIPTION:
Pre-operative anxiety is recognised as a potential and preventable risk factor for post-operative complications. It is estimated that between 25% to 80% of patients admitted to hospital for surgery experience pre-operative anxiety, and anxiety can negatively influence patient recovery.Physiologically pre-operative anxiety can lead to autonomic dysfunction and can modify inflammatory responses, platelet activity, and immunologic functioning. The Beck Anxiety Inventory(BAI), created by Aaron T. Beck is a 21 questions multiple choice self report inventory which measures the severity of an anxiety in adults and adolescents. It has been widely used in clinical research in mental health care mainly to measure general anxiety. The total score for all 21 symptoms can range between 0 and 63 points. A total score of 0 - 7 is interpreted as "Minimal" level of anxiety, 8 - 15 as "Mild"; 16 - 25 as "Moderate" and 26 - 63 as "Severe" level of anxiety.

This study aims to compare the alleviation of Pre-operative anxiety in patients undergoing surgery with or without music.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years scheduled for elective surgery
* American Society of Anaesthesiologists Physical Status I, II

Exclusion Criteria:

* Patient's refusal
* Patient's with known auditory disability
* Psychiatric disorder
* Altered mental status
* Patients routinely taking CNS depressant drugs (eg : Diazepam, Clonazepam)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
The effect of music therapy on preoperative anxiety in elective surgery | 6 months
  preoperative anxiety will be assessed by using Beck's Anxiety Inventory in one group and the other group will only get routine nursing care.The total score for all 21 symptoms can range between 0 and 63 points. A total score of 0 - 7 is interpreted as "Minimal" level of anxiety, 8 - 15 as "Mild"; 16 - 25 as "Moderate" and 26 - 63 as "Severe" level of anxiety. More the score greater the anxiety.

SECONDARY OUTCOMES:
The effect of music therapy on preoperative anxiety in elective surgery | 6 months
  systolic blood pressure
The effect of music therapy on preoperative anxiety in elective surgery | 6 months
  Diastolic blood pressure
The effect of music therapy on preoperative anxiety in elective surgery | 6 months
  mean arterial pressure
The effect of music therapy on preoperative anxiety in elective surgery | 6 months
  heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Anil Shrestha, MD, Study Director — TUTH; Bibhush Shrestha, MD, Study Director — MCVTC,IOM; Ninadini Shrestha, MD, Study Director — TUTH
Locations (1):
- Maharajgunj medical campus, TUTH, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stamenkovic DM, Rancic NK, Latas MB, Neskovic V, Rondovic GM, Wu JD, Cattano D. Preoperative anxiety and implications on postoperative recovery: what can we do to change our history. Minerva Anestesiol. 2018 Nov;84(11):1307-1317. doi: 10.23736/S0375-9393.18.12520-X. Epub 2018 Apr 5. PMID 29624026
- [Background] Tulloch I, Rubin JS. Assessment and Management of Preoperative Anxiety. J Voice. 2019 Sep;33(5):691-696. doi: 10.1016/j.jvoice.2018.02.008. Epub 2018 May 9. PMID 29753446
- [Background] Bae I, Lim HM, Hur MH, Lee M. Intra-operative music listening for anxiety, the BIS index, and the vital signs of patients undergoing regional anesthesia. Complement Ther Med. 2014 Apr;22(2):251-7. doi: 10.1016/j.ctim.2014.02.002. Epub 2014 Feb 23. PMID 24731896
- [Background] Lee WP, Wu PY, Lee MY, Ho LH, Shih WM. Music listening alleviates anxiety and physiological responses in patients receiving spinal anesthesia. Complement Ther Med. 2017 Apr;31:8-13. doi: 10.1016/j.ctim.2016.12.006. Epub 2017 Jan 7. PMID 28434475
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Lemos MF, Lemos-Neto SV, Barrucand L, Vercosa N, Tibirica E. [Preoperative education reduces preoperative anxiety in cancer patients undergoing surgery: Usefulness of the self-reported Beck anxiety inventory]. Braz J Anesthesiol. 2019 Jan-Feb;69(1):1-6. doi: 10.1016/j.bjan.2018.07.003. Epub 2018 Nov 3. PMID 30401475
- [Background] Franzoi MA, Goulart CB, Lara EO, Martins G. Music listening for anxiety relief in children in the preoperative period: a randomized clinical trial. Rev Lat Am Enfermagem. 2016 Dec 19;24:e2841. doi: 10.1590/1518-8345.1121.2841. PMID 27992027
- [Background] Jimenez-Jimenez M, Garcia-Escalona A, Martin-Lopez A, De Vera-Vera R, De Haro J. Intraoperative stress and anxiety reduction with music therapy: a controlled randomized clinical trial of efficacy and safety. J Vasc Nurs. 2013 Sep;31(3):101-6. doi: 10.1016/j.jvn.2012.10.002. PMID 23953858
- [Background] Wang Y, Dong Y, Li Y. Perioperative psychological and music interventions in elderly patients undergoing spinal anesthesia: effect on anxiety, heart rate variability, and postoperative pain. Yonsei Med J. 2014 Jul;55(4):1101-5. doi: 10.3349/ymj.2014.55.4.1101. PMID 24954343
- [Background] Ottaviani S, Bernard JL, Bardin T, Richette P. Effect of music on anxiety and pain during joint lavage for knee osteoarthritis. Clin Rheumatol. 2012 Mar;31(3):531-4. doi: 10.1007/s10067-011-1925-9. Epub 2011 Dec 30. PMID 22207250
- [Background] Ni CH, Tsai WH, Lee LM, Kao CC, Chen YC. Minimising preoperative anxiety with music for day surgery patients - a randomised clinical trial. J Clin Nurs. 2012 Mar;21(5-6):620-5. doi: 10.1111/j.1365-2702.2010.03466.x. Epub 2011 Feb 20. PMID 21332853
- [Background] Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: a report by the American Society of Anesthesiologist Task Force on Preoperative Fasting. Anesthesiology. 1999 Mar;90(3):896-905. doi: 10.1097/00000542-199903000-00034. No abstract available. PMID 10078693